CLINICAL TRIAL: NCT07330583
Title: Phase II Single Arm Study to Evaluate Stereotactic Body Radiation Therapy (SBRT) and Immunotherapy for Management of Patients With Oligometastatic Esophageal Cancer
Brief Title: Stereotactic Body Radiation Therapy (SBRT) and Immunotherapy for Oligometastatic Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0036
Record Dates: First submitted 2025-08-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT (Experimental)
  Interventions: Radiation: Stereotactic body radiation treatment (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiation treatment (SBRT) — Standard of care 6-9 cycles of chemotherapy and immunotherapy, which will then be followed by stereotactic body radiation treatment to the residual oligometastatic lesion/s.

SUMMARY:
Participants in this study will have esophageal cancer that has spread (metastasized) to other parts of the body either at initial diagnosis (synchronous) or after the cancer returned following treatment (recurrent).

In Alberta, the current standard approach for treating esophageal cancer that has metastasized is to first give patients radiation to the main tumor in the esophagus to relieve symptoms. After that, they receive a combination of chemotherapy drugs (either CAPOX or FOLFOX) chosen by their doctor, along with immunotherapy drugs like Pembrolizumab or Nivolumab to fight the cancer.

The study intends to add a treatment called stereotactic body radiation treatment (SBRT), which uses very high doses of radiation in a few sessions, to target small tumors which remain after the standard treatment.

The goal of this study is to see if adding SBRT to chemotherapy and immunotherapy helps patients with newly diagnosed or recurrent esophageal cancer that has metastasized to a few other places. The study aims to improve survival and control the disease better.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Eastern Cooperative Oncology Group performance status ≤ 2.
3. Histologically confirmed adenocarcinoma or squamous cell carcinoma of the esophagus.
4. Diagnosed with stage IVB disease (according to UICC TNM version 8) with up to five metastatic lesions in up to three organs.
5. At least one metastatic lesion amenable to the delivery of SBRT.
6. Estimated life expectancy >6 months.
7. The function of important organs meet the following requirements: a. white blood cell count (WBC) ≥ 4.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 100×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
8. Ability to understand the study and sign informed consent.
9. Women of childbearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
10. Patients of childbearing/reproductive potential should use highly effective birth control methods if indicated, as defined by the investigator, up to the period of finishing capecitabine and for 6 months after last dose. A highly effective method of birth control is defined as those that result in low failure rate (i.e., less than 1% per year) when used consistently and correctly. Note: abstinence is acceptable if this is established and preferred contraception for the patient.
11. Females must not be breastfeeding while taking capecitabine or within 2 weeks after the last dose.
12. Male patients should agree to not donate sperm during the study while taking capecitabine and for 3 months after the last dose.
13. Male patients should not father a child while taking capecitabine and for 3 months after the last dose.

Exclusion Criteria:

1. Progression was confirmed after completion of 4 to 6 cycles of standard chemotherapy and anti-PD1 treatment and not amenable to SBRT.
2. Known or suspected allergy or hypersensitivity to monoclonal antibodies and the chemotherapeutic drugs: Capecitabine, paclitaxel, or platinum.
3. Patients have spinal bone metastases combined with spinal cord compression.
4. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer.
5. Patients who cannot tolerate radiotherapy due to severe cardiac, lung, liver, or kidney dysfunction, or hematopoietic disease or cachexia.
6. Inability to provide informed consent due to psychological, familial, social, and other factors.
7. Female patients who are pregnant or during lactation.
8. Active autoimmune diseases, or a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism) that precludes the use of immunotherapy as decided by the treating medical oncologist, a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation.
9. A history of interstitial lung disease or non-infectious pneumonia; Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From the date of enrollment in the study for up to approximately 2 years and 7 months or death.
  Defined as time from enrollment into study to disease progression at any site or death.

SECONDARY OUTCOMES:
Local recurrence free survival | From the date of enrollment in the study for up to approximately 2 years and 7 months or death.
  Defined as time from enrollment into study to disease progression at site of SBRT treatment or death.
Overall Survival (OS) | From the date of enrollment until the time of death due to any cause, assessed up to approximately 2 years and 7 months
  Defined as the time from enrollment into study to death due to any cause.
Quality of Life (QOL) | Screening, 1 - 5 days before the start of each chemotherapy cycle (each cycle is 21 days), 14 - 28 days after completion of chemotherapy (chemotherapy is completed in about 4 months), and 3 monthly after SBRT until 2 years post SBRT
  To study the Quality of Life as measured by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) (v3)
Cancer Specific Survival (CSS) | From enrollment until the time of death due to esophageal cancer, assessed up to about 2 years and 7 months.
  Defined as the time from time of enrollment into study to death due to the esophageal cancer.
Toxicity Assessment | 10 - 20 days after screening (if given), 1 - 5 days prior each cycle of chemotherapy (each cycle is 21 days), 14 - 28 days after end of chemotherapy which is about 4 months, 14-28 days after chemotherapy and 3 monthly after SBRT until 2 years post SBRT.
  Treatment related toxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5

OTHER OUTCOMES:
To identify blood biomarkers that can correlate with disease events | Blood samples will be collected at baseline after signing consent, at time of completion of chemotherapy (chemotherapy takes 4 months), and 3 monthly after SBRT until 2 years post-SBRT.
  Blood samples will be compared between the baseline and subsequent samples for changes in the expression levels of specific markers that may be associated with metastases and treatment response. These include circulating cell free DNA and exosomes.